CLINICAL TRIAL: NCT00917553
Title: Proof-of-Concept 2 (POC2): Evaluation of Effect of Doxycycline Verses Placebo on Retinal Function and Diabetic Retinopathy Progression in Patients With Mild to Moderate Non-Proliferative Diabetic Retinopathy
Brief Title: Evaluation of Effect of Doxycycline Verses Placebo on Retinal Function and Diabetic Retinopathy
Acronym: POC2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Thomas Gardner (Other)
Collaborators: Penn State University (Other); Juvenile Diabetes Research Foundation (Other)
Responsible Party: Sponsor-Investigator, Thomas Gardner, Thomas W. Gardner, MD, Milton S. Hershey Medical Center
Organization: Milton S. Hershey Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 30791
Record Dates: First submitted 2009-06-01; First posted 2009-06-10 (Estimated); Results first posted 2018-11-30 (Actual); Last update posted 2018-11-30 (Actual); Status verified 2018-10

CONDITIONS: Diabetic Retinopathy
Keywords: diabetic retinopathy; diabetes; diabetic eye studies
MeSH Terms: conditions — Diabetic Retinopathy; Diabetes Mellitus | interventions — Doxycycline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- doxycycline monohydrate (Experimental)
  Interventions: Drug: doxycycline monohydrate
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: doxycycline monohydrate — 50 mg
  Arms: doxycycline monohydrate
Drug: Placebo — Cellulose Placebo Capsule
  Arms: Placebo

SUMMARY:
This 24 month randomized research study will evaluate whether doxycycline can slow the deterioration or improve retinal function among patients with mild to moderate non-proliferative diabetic retinopathy.

DETAILED DESCRIPTION:
The objective of this proof-of-concept study is to investigate whether doxycycline can slow the deterioration or improve retinal function among patients with mild to moderate NPDR (with abnormal retinal function defined as a foveal sensitivity < 30.91 dB on Matrix frequency doubling perimetry [FDP]). Based on results of the END DR Study, the primary visual function endpoint in the POC 2 Study will be performance on the Matrix Frequency Doubling Technology Perimeter. This test was the most sensitive to NPDR of the visual function endpoints the investigators evaluated in the END DR Study. This selection is aggressive because the investigators lack natural history data to estimate the 2-year rate of change in the endpoint; in fact, a major output of this POC 2 Study will be 2-year natural history data using several visual function endpoints. The investigators are enrolling patients who have moderate dysfunction; that is, patients who fall outside the 95% confidence interval of normal performance on FDP. These patients will have the opportunity to improve their FDP performance to "normal" levels as well as progress to more severe FDP impairment associated with more advanced disease. Secondary endpoints include visual acuity, contrast sensitivity, visual field, and dark adaptation. The tests will be performed in the Ophthalmology Department of the Penn State College of Medicine. The 24-month proof-of-concept clinical study will involve a prospective, randomized, double-masked clinical trial including 60 adult patients with type 1 or type 2 diabetes who have mild to moderate NPDR (ETDRS levels 20 to 43), and in whom retinal photocoagulation is not anticipated (by the investigator) within the subsequent 2 years. Participants will be randomized to receive either doxycycline monohydrate 50mg or an identical placebo once daily for 24 months.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years old
* diagnosis of type 1 or type 2 diabetes mellitus (defined as current regular use of oral anti-hyperglycemia agents and/or insulin for the treatment of diabetes)
* have a hemoglobin A1c < 11% at pre-qualification visit
* able and willing to give informed consent
* best-corrected ETDRS visual acuity (10) in study eye ≥ 69 letters (20/40)
* mild to moderate non-proliferative diabetic retinopathy (ETDRS levels 20 to 43) (11), and in whom retinal photocoagulation is not anticipated (by the investigator) within the subsequent 2 years
* able to perform reliable visual field and dark adaptation testing
* central subfield thickness on OCT ≤ 275 microns
* media clarity and pupil dilation sufficient for high-quality fundus photographs
* abnormal retinal function defined as:
* abnormal FDP function as defined by a foveal sensitivity ≤ 30.91 dB

Exclusion Criteria:

* prior panretinal photocoagulation in the study eye
* prior focal/grid laser photocoagulation in the macula in the study eye
* intraocular pressure in the study eye > 22 mmHg by Goldmann tonometry
* history of pars plana vitrectomy in the study eye
* systemic or intravitreal anti-VEGF agent to the study eye or the fellow eye within the past 3 months
* peribulbar steroid injection to the study eye or the fellow eye within the past 6 months
* intravitreal triamcinolone acetonide to the study eye within the past 4 months
* expectation by the investigator that retinal photocoagulation or other treatment for diabetic retinopathy (e.g., focal/grid laser to study eye, intravitreal triamcinolone acetonide to study eye, intravitreal anti-VEGF agent to study or fellow eye, ruboxistaurin or systemic anti-VEGF agent for diabetic macular edema) will be administered in the subsequent 24months
* an ocular condition (other than diabetes) is present in the study eye that, in the opinion of the investigator, might alter visual acuity during the course of the study (e.g., retinal vein occlusion, uveitis or other ocular inflammatory disease, neovascular glaucoma, Irvine-Gass Syndrome, etc)
* anticipated need for cataract surgery in the study eye in the subsequent 24 months in the opinion of the investigator
* history of major ocular surgery (including cataract surgery, scleral buckle, any intraocular surgery, etc) in the study eye within prior 6 months or anticipated within the subsequent 24 months following randomization
* aphakia in the study eye
* history of YAG capsulotomy performed in the study eye within 2 months prior to randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2009-07; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas W Gardner, MD.,MS., Study Director — University of Michigan, Kellogg Eye Center
Locations (1):
- Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

REFERENCES:
- [Derived] Scott IU, Jackson GR, Quillen DA, Klein R, Liao J, Gardner TW. Effect of doxycycline vs placebo on retinal function and diabetic retinopathy progression in mild to moderate nonproliferative diabetic retinopathy: a randomized proof-of-concept clinical trial. JAMA Ophthalmol. 2014 Sep;132(9):1137-42. doi: 10.1001/jamaophthalmol.2014.1422. PMID 24969516

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Doxycycline Monohydrate
Started | 17 | 16
Completed | 15 | 15
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Doxycycline Monohydrate | Total
Number analyzed (Participants) | 17 | 16 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.76 (7.61) | 58.44 (12.96) | 57.57 (10.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 12 | 9 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 17 | 15 | 32
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 17 | 16 | 33

OUTCOME MEASURES:

1. Primary Outcome: The Mean Change in the Foveal Sensitivity of Matrix Frequency Doubling Perimetry (FDP) From Baseline in the Treated Group Compared to the Placebo Group
Time Frame: Baseline and 24 months
Population: Two participants in the placebo group and one in the doxycycline group were unavailable for 24 month results.
Measure: Mean (Standard Deviation); unit: dB
Arm/Group | Placebo | Doxycycline Monohydrate
Number analyzed (Participants) | 15 | 15
dB | 2.80 (3.80) | 0.13 (4.45)

2. Secondary Outcome: Change Thickness Thickness
Description: Anatomic outcomes were assessed through optical coherence. Positive numbers indicate increases in thickness.
Time Frame: Baseline and 24 months
Measure: Mean (Standard Deviation); unit: µm
Arm/Group | Placebo | Doxycycline Monohydrate
Number analyzed (Participants) | 15 | 15
µm
  Central subfield thickness | 17.5 (27.3) | 21.3 (72.5)
  Center point thickness | 25.6 (41.7) | 26.1 (81.1)

3. Secondary Outcome: Change in Macular Volume
Time Frame: Baseline and 24 months
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | Placebo | Doxycycline Monohydrate
Number analyzed (Participants) | 15 | 15
mm^3 | 0.06 (0.34) | 0.23 (0.67)

4. Secondary Outcome: Number of Participants With Progression to PDR, and Single or Multiple Step Progression in ETDRS Diabetic Retinopathy Severity Level
Description: Participants are shown categorically by whether they reached PDR, or whether their diabetic retinopathy levels changed by one grade or more, as analyzed by fundus photography.
Time Frame: Baseline to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Doxycycline Monohydrate
Number analyzed (Participants) | 17 | 16
Participants
  Progressed to PDR | 0 | 1
  >=1 severity level ETDRS | 9 | 7
  >=2 severity level ETDRS | 0 | 2
  >=3 severity level ETDRS | 0 | 1

5. Secondary Outcome: Number of Participants Who Developed Vitreous or Preretinal Hemorrhage
Description: Any participants who developed vitreous or preretinal hemorrhage were counted. Had there been any preretinal hemorrhages (a subcategory of vitreous hemorrhage) these would have been shown as a separate row.
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Doxycycline Monohydrate
Number analyzed (Participants) | 15 | 15
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | Placebo | Doxycycline Monohydrate
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/16
Serious Adverse Events (participants affected / at risk) | 4/17 | 8/16
Other Adverse Events (participants affected / at risk) | 16/17 | 14/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=17) | Doxycycline Monohydrate (N=16)
dysphagia (Musculoskeletal and connective tissue disorders) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 1
E. Coli sepsis/acute kidney injury (Infections and infestations) | 1 | 0
probable TIA (Cardiac disorders) | 1 | 0
arthritis - total knee arthroplasty (Musculoskeletal and connective tissue disorders) | 0 | 1
diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 1
angina/non-anginal chest pain (Cardiac disorders) | 1 | 0
hospitalization - noncardiac chest pain (General disorders) | 1 | 0
chronic renal failure (Renal and urinary disorders) | 0 | 1
confusional state (Psychiatric disorders) | 0 | 1
uncontrolled hyperglycemia (Metabolism and nutrition disorders) | 2 | 0
chronic systolic heart failure (Cardiac disorders) | 0 | 1
right foot Charcot arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Mobitz type 1 (Cardiac disorders) | 1 | 0
accelerated hypertension (Cardiac disorders) | 1 | 0
unstable angina (Cardiac disorders) | 1 | 0
acute bronchitis requiring hospitalization (Respiratory, thoracic and mediastinal disorders) | 1 | 0
possible seizure with hospitalization (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=17) | Doxycycline Monohydrate (N=16)
glaucoma (Eye disorders) | 0 | 1
4 broken toes left foot (Musculoskeletal and connective tissue disorders) | 0 | 1
acid reflux (Gastrointestinal disorders) | 2 | 0
arm weakness and numbness (Musculoskeletal and connective tissue disorders) | 1 | 0
arthritis (Musculoskeletal and connective tissue disorders) | 0 | 2
bilateral excision of ingrown toenails of big toes (Surgical and medical procedures) | 0 | 1
bloating (Gastrointestinal disorders) | 1 | 0
blood in urine / kidney stone (Renal and urinary disorders) | 1 | 0
blurry vision (Eye disorders) | 2 | 1
bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
bursitis left knee (Musculoskeletal and connective tissue disorders) | 0 | 1
cellulitis left leg (Infections and infestations) | 1 | 0
Charcot right foot and ankle (Nervous system disorders) | 1 | 0
back pain (Musculoskeletal and connective tissue disorders) | 1 | 3
cloudy left eye (Eye disorders) | 0 | 1
chest cold (Respiratory, thoracic and mediastinal disorders) | 2 | 4
intestinal flu (Gastrointestinal disorders) | 0 | 1
shoulder pain (Musculoskeletal and connective tissue disorders) | 1 | 1
macular edema (Eye disorders) | 0 | 1
dehydration (General disorders) | 0 | 1
depression (Psychiatric disorders) | 2 | 2
dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
diarrhea (Gastrointestinal disorders) | 1 | 1
diplopia (Eye disorders) | 0 | 1
dry eyes (Eye disorders) | 0 | 1
episodal gout (Metabolism and nutrition disorders) | 1 | 0
fluid retention (Renal and urinary disorders) | 1 | 0
gum infection (Infections and infestations) | 0 | 1
herniated nucleus pulposus (Musculoskeletal and connective tissue disorders) | 1 | 0
high calcium (Metabolism and nutrition disorders) | 0 | 1
hives (Immune system disorders) | 2 | 0
hypertension (Cardiac disorders) | 1 | 1
ingrown hair left forearm (Skin and subcutaneous tissue disorders) | 1 | 0
hip pain (Musculoskeletal and connective tissue disorders) | 1 | 0
joint pain (Musculoskeletal and connective tissue disorders) | 1 | 0
kidney stone (Renal and urinary disorders) | 1 | 0
systemic capillary leak syndrome (Blood and lymphatic system disorders) | 1 | 0
MRSA (Infections and infestations) | 1 | 0
muscle aches (Musculoskeletal and connective tissue disorders) | 1 | 0
muscle spasms over heart (Musculoskeletal and connective tissue disorders) | 1 | 0
nausea (Gastrointestinal disorders) | 1 | 1
neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
ocular migraine (Eye disorders) | 1 | 0
posterior capsule opacification (Eye disorders) | 1 | 0
peripheral neuropathy (Nervous system disorders) | 2 | 0
possible broken left thumb (Musculoskeletal and connective tissue disorders) | 1 | 0
probable seizure (Nervous system disorders) | 0 | 1
right eye corneal abrasion (Eye disorders) | 0 | 1
right foot plantar fascitis (Musculoskeletal and connective tissue disorders) | 1 | 0
right heel pain (Musculoskeletal and connective tissue disorders) | 1 | 0
right knee pain (Musculoskeletal and connective tissue disorders) | 0 | 1
right rotator cuff tear (Musculoskeletal and connective tissue disorders) | 1 | 0
seasonal allergies (Immune system disorders) | 1 | 0
sinus infection (Respiratory, thoracic and mediastinal disorders) | 2 | 1
sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
sleep trouble (General disorders) | 0 | 1
stenosis tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 | 0
strain to left knee ligaments and tendons (Musculoskeletal and connective tissue disorders) | 1 | 0
tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0
trouble breathing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
urinary tract infection (Renal and urinary disorders) | 1 | 1
right foot infection (Infections and infestations) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No